CLINICAL TRIAL: NCT05209620
Title: A Single Arm, Phase II Clinical Trial of Orelabrutinib Combined With Pemetrexed in the Treatment for Patients With Relapsed/Refractory Central Nervous System Lymphoma
Brief Title: Orelabrutinib Combined With Pemetrexed For Relapsed/Refractory Central Nervous System Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhihua Yao, PhD, Director, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNSZLYYNHL06
Record Dates: First submitted 2021-12-26; First posted 2022-01-26 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Central Nervous System Lymphoma
Keywords: Central Nervous System Lymphoma; BTK inhibitor; Relapsed and Refractory
MeSH Terms: conditions — Recurrence | interventions — orelabrutinib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Orelabrutinib Combined with Pemetrexed (Experimental): Induction Chemotherapy: Orelabrutinib, 150mg/d continuous oral administration, Pemetrexed, 500mg/m2, Intravenous administration on day 5 of each 3-week cycle (Total 6 cycles).
  Maintenance Treatment: Orelabrutinib, 150mg/d continuous oral administration (28d/cycle).
  Interventions: Drug: ICP-022; Drug: Pemetrexed

INTERVENTIONS:
Drug: ICP-022 — Induction Chemotherapy: Orelabrutinib, 150mg/d continuous oral administration (3 weeks/cycle, total 6 cycles).
  Maintenance Treatment: Orelabrutinib, 150mg/d continuous oral administration (28d/cycle).
  Other Names: orelabrutinib
Drug: Pemetrexed — Induction Chemotherapy: Pemetrexed, 500mg/m2, Intravenous administration on day 5 of each 3-week cycle (Total 6 cycles).
  Other Names: Pemetrexed injection

SUMMARY:
This is a prospective single arm, phase II clinical trial to observe the efficacy and safety of orelabrutinib combined with pemetrexed in the treatment for patients with relapsed/refractory central nervous system lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 75 years old (including 18 and 75)
2. Diagnosed as diffuse large B-cell lymphoma; Recurrence or progression of central nervous system disease confirmed by imaging ± tissue biopsy pathology or cerebrospinal fluid flow cytometry; Secondary central nervous system lymphoma can also be admitted when the systemic disease is well controlled
3. Having at least one measurable lesions
4. World health organization-Eastern Cooperative Oncology Group Performance Status (ECOG) 0-2 ( ECOG 3 due to tumors can be included after being fully assessed by the investigator)
5. Life expectancy no less than 1 month
6. enough main organ function
7. Pregnancy test within 7 days must be negative for women of childbearing period, and appropriate measures should be taken for contraception for women in childbearing period during the study and six months after this study
8. Agreeing to sign the written informed consents

Exclusion Criteria:

1. Poor peripheral disease control of secondary central nervous system lymphoma
2. Patients used pemetrexed or orelabrutinib in the past
3. Active malignant tumor need be treated at the same time
4. Other malignant tumor history
5. Serious surgery and trauma less than two weeks
6. Patients with active tuberculosis
7. Systemic therapy for serious acute/chronic infection
8. Congestive heart failure, uncontrolled coronary heart disease, arrhythmia and heart infarction less than 6 months
9. HIV-positive, AIDS patients and untreated active hepatitis
10. Patients with a history of deep vein thrombosis or pulmonary embolism less than 12 months
11. Patients with a history of mental illness or drug abuse
12. Poor compliance during the trial and/or follow-up phase
13. Allergies or people who are known to be allergic to any active ingredients, excipients, mouse-derived products or heterologous protein contained in this trial
14. Researchers determine unsuited to participate in this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
objective response rate | every 6 weeks from the day of the first cycle of induction chemotherapy treatment (each cycle is 21 days) and every 8 weeks from the day of the first cycle of maintenance treatment to 5 years after last patient's enrollment (each cycle is 28 days)
  the total proportion of patients with complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
progression-free survival | every 6 weeks from the day of the first cycle of induction chemotherapy treatment (each cycle is 21 days) and every 8 weeks from the day of the first cycle of maintenance treatment to 5 years after last patient's enrollment (each cycle is 28 days)
  the total proportion of patients with no progression from date of the first day of treatment to the date of confirmed progressive disease or death which one occurs first
overall survival | every 6 weeks from the day of the first cycle of induction chemotherapy treatment (each cycle is 21 days) and every 8 weeks from the day of the first cycle of maintenance treatment to 5 years after last patient's enrollment (each cycle is 28 days)
  from date of first day of treatment to the date of death by any cause
The incidence of grade 3-4 adverse events | up to 5 years
  the incidence of grade 3 or 4 adverse events (based on NCI CTC-AE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Zhihua Yao, M.D. Ph.D, Study Director — Henan Cancer Hospital; Yanyan Liu, M.D. Ph.D, Study Director — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No